CLINICAL TRIAL: NCT05611632
Title: A Randomized, Controlled Trial to Assess the Clinical Utility of a Multi-cancer Early Detection (MCED) Test for Population Screening in the United Kingdom (UK) When Added to Standard of Care
Brief Title: Does Screening With the Galleri Test in the NHS Reduce the Likelihood of a Late-stage Cancer Diagnosis in an Asymptomatic Population? A Randomised Clinical Trial
Acronym: NHS-Galleri
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GRAIL, Inc. (Industry)
Collaborators: The Cancer Research UK Cancer Prevention Trials Unit at Queen Mary University of London (CPTU) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: GRAIL-009; ISRCTN91431511 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2022-10-28; First posted 2022-11-10 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: multi-cancer early detection; cancer screening; MCED; circulating cell-free tumor DNA
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to either the intervention arm, with blood collection and evaluation of the test with consequent investigation and treatment of a positive test through referral to the NHS urgent two week wait pathway, or to the control arm, where blood samples are collected at designated intervals and will be stored for potential future evaluation, but participants do not receive test results and otherwise continue to receive routine NHS care.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Interventional (Experimental): Blood collection and multi-cancer early detection testing with return of positive test results.
  Interventions: Device: Multi-cancer early detection test (Galleri test)
- Control (No Intervention): Blood collection only.

INTERVENTIONS:
Device: Multi-cancer early detection test (Galleri test) — Blood collection and multi cancer early detection testing with return of positive test results.
  Other Names: Galleri test
  Arms: Interventional

SUMMARY:
The Galleri test is a new test that looks for potential signs of cancer in a blood sample. The test can find many different types of cancer but cannot find all cancers. The trial aims to see if using the Galleri test alongside standard cancer testing in the NHS can help to find cancers at an early stage when they are easier to treat.

The trial has enrolled approximately 140,000 participants who will be actively followed for approximately three years from the date of enrollment.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled trial to assess the performance and clinical utility of a multi-cancer early detection test for population screening in the UK when added to standard of care. Participants and the study teams remain blinded throughout the study with the exception of the study nurses returning the results and a small number of staff to enable them to perform administrative duties. Blinding is maintained for participants with the exception of those participants who test positive. Those who test positive will be informed by designated trial staff and will be referred for standard of care investigations and treatment. Trial sponsor employees, the CIs and site staff (unless identified differently in the blinding plan for study conduct needs) will remain blinded throughout the study.

Randomization will be to either the intervention arm, with blood collection and evaluation of the test with consequent investigation and treatment of a positive test through referral to the NHS urgent two week wait pathway, or to the control arm, where blood samples are collected at designated intervals and will be stored for potential future evaluation, but participants do not receive test results and otherwise continue to receive routine NHS care.

Unless diagnosed with cancer, participants in both arms will be asked to return for annual visits at approximately 12 and 24 months. All participants whether test positive, test negative or not tested will be followed for cancer and associated outcomes via NHS dataset linkages.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be at 50-77 years of age, inclusive, at the time of data extraction from NHS datasets or GP records used to identify potential participants; and
2. Capable of giving signed and legally effective informed consent, which includes compliance with the requirements and restrictions listed in the Informed Consent Form (ICF) and in this protocol. Consent provided by a legally authorised representative is not permitted in this protocol.

Exclusion Criteria:

1. Previous or current participation in another GRAIL-sponsored study.
2. Personal history of invasive cancer or haematologic malignancy, diagnosed within the three years prior to expected enrolment date. Note: Individuals with a diagnosis of non-melanoma skin cancer and prostate cancer patients whose only treatment is active surveillance are NOT excluded
3. Definitive treatment for invasive cancer or haematologic malignancy within the 3 years prior to expected enrolment date, including adjuvant hormone therapy for cancer (e.g. for breast or prostate cancer).
4. Currently taking demethylating or cytotoxic agents for any condition.
5. Undergoing current investigation for suspected cancer, defined as having been referred to a two week wait clinic or undergoing investigations at an RDC or other clinic with a stated suspicion of cancer.
6. Currently on a palliative care pathway.

Ages: 50 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142318 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
absolute numbers of stage III and IV cancers diagnosed | 3-4 years after randomization

SECONDARY OUTCOMES:
absolute numbers of advanced cancers (stage III and IV cancers or one that results in a cancer-specific death) diagnosed | 3-4 years after randomization
absolute numbers of stage IV cancers diagnosed | 1 years after randomization
absolute numbers of stage IV cancers diagnosed | 3-4 years after randomization
cancer-specific mortality | up to 8 years after randomization
proportion of Stage I and II cancers | 3-4 years after randomization
test performance (sensitivity, specificity, positive predictive value, negative predictive value) and cancer signal origin accuracy) in the intervention arm. | Up to 3 years
number of follow up procedures and invasive procedures, complications and deaths associated with follow-up diagnostic procedures in all test positive cases | Up to 3 years
number and type of invasive procedures performed in false positive cases | Up to 3 years
radiation exposure measured in mSv per participant due to test result directed evaluations in all test positive cases | Up to 3 years
psychological impact using the short form State Trait Anxiety Index-6 questionnaire (a six item validated measure of state anxiety), at various timepoints in all test positive cases | Up to 3 years
  Scores range from 20-80 with the general population expected to score 34-36 and very high anxiety classed as scoring > 49.

OTHER OUTCOMES:
healthcare resource utilisation | Up to 3 years
  The data collected may be used to conduct future exploratory economic analyses, and will include: Number and types of medical encounters and cancer-specific diagnostic and treatment procedures, including clinical lab visits, imaging tests, invasive tests, and clinic visits.

CONTACTS AND LOCATIONS:
Overall Officials: Poorwa Roy, Study Director — GRAIL, Inc.
Locations (1):
- EMS Healthcare Ltd, Chester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marlow LAV, Schmeising-Barnes N, Warwick J, Waller J. Psychological Impact of the Galleri test (sIG(n)al): protocol for a longitudinal evaluation of the psychological impact of receiving a cancer signal in the NHS-Galleri trial. BMJ Open. 2023 Jul 21;13(7):e072657. doi: 10.1136/bmjopen-2023-072657. PMID 37479515
- [Background] Neal RD, Johnson P, Clarke CA, Hamilton SA, Zhang N, Kumar H, Swanton C, Sasieni P. Cell-Free DNA-Based Multi-Cancer Early Detection Test in an Asymptomatic Screening Population (NHS-Galleri): Design of a Pragmatic, Prospective Randomised Controlled Trial. Cancers (Basel). 2022 Oct 1;14(19):4818. doi: 10.3390/cancers14194818. PMID 36230741
- [Background] Brentnall AR, Mathews C, Beare S, Ching J, Sleeth M, Sasieni P. Dynamic data-enabled stratified sampling for trial invitations with application in NHS-Galleri. Clin Trials. 2023 Aug;20(4):425-433. doi: 10.1177/17407745231167369. Epub 2023 Apr 24. PMID 37095697
- [Derived] Marlow LAV, Schmeising-Barnes N, Waller J. Experience of NHS diagnostic investigation following a multi-cancer early detection (MCED) screening test: qualitative interviews with NHS-Galleri trial participants who had a cancer signal detected. EClinicalMedicine. 2026 Jan 8;91:103733. doi: 10.1016/j.eclinm.2025.103733. eCollection 2026 Jan. PMID 41567711
- [Derived] Swanton C, Bachtiar V, Mathews C, Brentnall AR, Lowenhoff I, Waller J, Bomb M, McPhail S, Pinches H, Smittenaar R, Hiom S, Neal RD, Sasieni P. NHS-Galleri trial: Enriched enrolment approaches and sociodemographic characteristics of enrolled participants. Clin Trials. 2025 Apr;22(2):227-238. doi: 10.1177/17407745241302477. Epub 2025 Jan 25. PMID 39862108
- [Derived] Smittenaar R, Quaife SL, von Wagner C, Higgins T, Hubbell E, Lee L. Impact of screening participation on modelled mortality benefits of a multi-cancer early detection test by socioeconomic group in England. J Epidemiol Community Health. 2024 May 9;78(6):345-353. doi: 10.1136/jech-2023-220834. PMID 38429085